CLINICAL TRIAL: NCT05736419
Title: Pre-Transplant Immune Suppression With Hematopoietic Cell Transplantation From Haploidentical Donors for Adults and Children With Sickle Cell Disease or ß-Thalassemia (Haplo PTCy)
Brief Title: A Study of Immune Suppression Treatment for People With Sickle Cell Disease or β-Thalassemia Who Are Going to Receive an Allogeneic Hematopoietic Cell Transplantation (HCT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-009
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease; Thalassemia, Beta; Thalassemia
Keywords: allogeneic hematopoietic cell transplantation; Sickle Cell Disease; Beta Thalassemia; Thalassemia; 23-009; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia; Thalassemia | interventions — fludarabine; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; thymoglobulin; Dexamethasone; Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Sickle Cell Disease or β-Thalassemia (Experimental): Participants will have severe sickle cell disease or transfusion-dependent β-thalassemia.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Biological: Rabbit ATG; Drug: Dexamethasone; Drug: Bortezomib; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine — PK-guided fludarabine dosing will be used for each of the 2 cycles, using the InsightRx DoseMeRx platform.
Drug: Cyclophosphamide — Cyclophosphamide will be administered Post-Transplant
Drug: Tacrolimus — Tacrolimus will be administered beginning on day +5
Drug: Mycophenolate Mofetil — Mycophenolate mofetil (MMF) will be administered three times daily starting on day +5.
Biological: Rabbit ATG — The dose and schedule of ATG will be determined according to the nomogram in Appendix A
Drug: Dexamethasone — Standard Regimen: Dexamethasone on days -68 to -64 and days -40 to -36.
Drug: Bortezomib — Bortezomib on days -71, -68, -65, -61, -43, -40, -37, and -33
Drug: Rituximab — Rituximab on days -71, -58, -43, and -30.

SUMMARY:
Hematopoietic Cell Transplantation/HCT involves receiving healthy blood-forming cells (stem cells) from a donor to replace the diseased or damaged cells in participants' bone marrow. The researchers think giving participants treatment with fludarabine and dexamethasone, drugs that lower the activity of the body's immune system (immune suppression), before standard conditioning therapy and HCT may help prevent serious side effects, including graft failure and GvHD. In this study, depending on how participants' body responds to the fludarabine and dexamethasone, the study doctor may decide participants should receive another drug, called cyclophosphamide, instead of fludarabine. In addition, depending on the results of participants' routine blood tests, participants may receive the drugs bortezomib and rituximab, which also help with immune suppression.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 and < 35 years. Patients of age 2-12 and 35-50 years will be included after 8 patients reach day 100 without TRM and if ≥ 4 of the first 8 patients reach day 100 without graft failure or grade III-IV acute GvHD.
* Suitable haploidentical donor.
* Performance score ≥ 70% by Karnofsky Performance Scale or 0 to 1 by ECOG (age > 16 years), or Lansky Play-Performance Scale ≥ 70% (age ≤ 16 years).
* Adequate major organ system function as demonstrated by:

  * For patients ≥ 18 years of age:
  * eGFR ≥ 50 mL/min by Cockcroft-Gault formula
  * For patients < 18 years of age:
  * Serum creatinine clearance: glomerular filtration rate [GFR]) must be >50 mL/min/1.73 m2 as calculated by the Schwartz formula
* Conjugated (direct) bilirubin less than 2x upper limit of normal.
* ALT or AST ≤ 3 times institutional upper limit of normal.
* Left ventricular ejection fraction ≥ 50%.
* Diffusing capacity for carbon monoxide (DLCO) ≥ 50% predicted, corrected for hemoglobin. For children < 7 years of age who are unable to perform PFT, oxygen saturation > 92% on room air by pulse oximetry.
* For SCD patients: HbSS, HbSC, HbS/β° with one or more of the following complications:

  * Acute chest syndrome: 2 or more episodes in the 2 years preceding enrollment
  * Vaso-occlusive episodes: 3 or more episodes in the 2 years preceding enrollment
  * Recurrent priapism: 2 or more episodes in the 2 years preceding enrollment
  * History of osteomyelitis or osteonecrosis
  * Cerebrovascular disease:
* Imaging evidence of prior overt or silent stroke
* History of a neurologic event resulting in focal neurologic deficits lasting > 24 hours
* Abnormal transcranial Doppler: Timed average maximum mean velocity ≥ 200 cm/sec in terminal portion of the carotid or proximal portion of the middle cerebral artery or > 185 cm/sec plus evidence of intracranial vasculopathy if imaging TCD is used

  * Pulmonary hypertension: Confirmed by right heart catheterization with mean pulmonary arterial pressure ≥ 25 mmHg or mean pulmonary vascular resistance > 2 Wood units
  * Red blood cell alloimmunization (> 3 alloantibodies)
* For thalassemia patients: Any genotype, with all of the following:

  * Onset of red blood cell transfusion dependence during the first 3 years of life
  * RBC transfusion history > 225 mL/kg/year or > 15 lifetime RBC transfusions
  * Pre-transfusion hemoglobin ≤ 7 g/dL
  * Hepatosplenomegaly
* Patient or the patient's legal representative, parent(s) or guardian should be able to provide written informed consent. Assent of a minor if participant's age is at least seven and less than eighteen years.
* For sexually active men and women of childbearing potential, must agree to use a form of contraception considered effective and medically acceptable by the Investigator.

Exclusion Criteria:

* Prior myeloablative allogeneic HCT.
* Overt stroke or CNS instrumentation (e.g. for Moyamoya disease) within 6 months of enrollment.
* Liver cirrhosis. Mild fibrosis will be permitted, i.e. fine reticulin or grade 1 of 4, with bridging fibrosis.
* Hepatic iron content ≥ 3 mg Fe/g liver dry weight
* HIV positive
* Active hepatitis B or C.
* Other uncontrolled infections.
* BMI > 40.
* Other malignancy/cancer diagnosis unless in remission after definitive therapy for a minimum of 2 years. Exceptions: Ductal carcinoma in situ, basal cell carcinoma, cervical intraepithelial neoplasia.
* Positive pregnancy test in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization.
* Inability to comply with medical therapy or follow-up.
* Known history of allergic reactions to any constituents of the cell product, including a known history of allergic reactions to DMSO.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related mortality/TRM or primary graft failure | 1 year
  The primary outcome is to estimate treatment-related mortality (TRM) or primary graft failure at 1 year post-HCT.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cancio, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org